CLINICAL TRIAL: NCT06876584
Title: The CT-based Deep Learning Model Outperforms Traditional Anatomical Classification Models in Preoperatively Predicting Complications and Risk Grade in Partial Nephrectomy
Brief Title: The CT-based Deep Learning Model Predicts Complications in Partial Nephrectomy
Status: Completed | Type: Observational
Sponsor: Du Lingzhi (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Minhang Hospital, Fudan University (Unknown); Xuhui Central Hospital, Shanghai (Other)
Responsible Party: Sponsor-Investigator, Du Lingzhi, Principal Investigator, Fudan University
Organization: Fudan University (Other)
Other Study IDs: zsurologyDLMforPNcomplication
Record Dates: First submitted 2025-03-08; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Renal Cell Carcinoma (RCC); Renal Cyst
Keywords: CT-based deep learning; complication prediction; traditional classification model; partial nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Complication 1: Patients who experienced perioperative complications during the partial nephrectomy
- Complication 0: Patients who didn't experience perioperative complications during the partial nephrectomy

SUMMARY:
The investigators combine radiomics and deep learning to analyze the lesions more thoroughly, aiming for a more accurate prediction of complications in partial nephrectomy, and compare this approach with traditional models.

DETAILED DESCRIPTION:
In this study, patients diagnosed with renal cell carcinoma or renal cyst who underwent partial nephrectomy across multiple centers was included. And the participants were excluded if they had (a) missing or unavailable imaging data or (b) no available enhanced CT images. The cohort was divided into training and test sets at a 7:3 ratio. After that, the radiomics features were extracted from the images, and lasso regression was used to select features. Then a deep learning model was developed to predict complications and risk grades and compared with traditional classification models (RENAL and PADUA), demonstrating superior applicability.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of renal cell carcinoma or renal cyst
* Underwent partial nephrectomy between June 2014 and July 2024

Exclusion Criteria:

* Missing or unavailable imaging data
* No available enhanced CT images

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes patients diagnosed with renal cell carcinoma or renal cyst who underwent partial nephrectomy in the participated centers. Clinical and imaging data were retrospectively collected from medical records, including demographic characteristics (age, gender, BMI), tumor location (left or right kidney), surgical details (surgical approach, ischemia time), and perioperative complications.
  Patients were included based on the availability of complete clinical, surgical, and imaging data. Exclusion criteria comprised individuals with missing or unavailable imaging data, or no available enhanced CT images. The study aims to combine CT-based radiomics features and clinical features to develop a deep learning model to predict perioperative complications of partial nephrectomy, and compare with traditional anatomical classification models.
Sampling Method: Non-Probability Sample
Enrollment: 1474 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
whether complications occurred | perioperatively
  Retrospectively review the medical record system to determine whether patients developed postoperative complications.

SECONDARY OUTCOMES:
Patients' risk grade | perioperatively
  Based on the widely recognized Clavien-Dindo classification (CDC) system for surgical complications, these complications were categorized into four grades: Grade I, II, III, and IV. Risk grade was assigned accordingly: "no risk" is defined as no complications occurred, "grade low" is defined as the highest level of complication being Grade I, "grade moderate" is defined as the highest level of complication being Grade II, and "grade high" is defined as complications of Grade III or higher, which are life-threatening.

CONTACTS AND LOCATIONS:
Locations (1):
- Name: Zhongshan Hospital Fudan University, Location: 180th Fenglin Road, Xuhui District, Shanghai, China, Shanghai, Xuhui District, China

IPD SHARING:
Plan to Share IPD: Yes
Clinical data and extracted radiomics feature data, excluding patient information.
Supporting Information: Study Protocol
Time Frame: Within six months after publication in the journal.
Access Criteria: The data supporting this study are available from the enrolled institutions, but restrictions apply to their availability due to privacy reasons. Data can be accessed upon reasonable request from the corresponding author.